CLINICAL TRIAL: NCT06148051
Title: AusCADASIL: An Australian Cohort of CADASIL
Status: Recruiting | Type: Observational
Sponsor: Perminder Sachdev (Other)
Collaborators: Prince of Wales Hospital, Sydney (Other Government); John Hunter Hospital (Other Government); St Vincent's Hospital - Sydney, Australia (Other); Royal Brisbane and Women's Hospital (Other Government); Melbourne Health (Other); The University of Queensland (Other)
Responsible Party: Sponsor-Investigator, Perminder Sachdev, Professor, The University of New South Wales
Organization: The University of New South Wales (Other)
Other Study IDs: AusCADASIL
Record Dates: First submitted 2023-11-07; First posted 2023-11-28 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Cadasil
Keywords: CADASIL; Clinical Research; Genetics; Cognition; Neuroimaging; Blood markers; Retinal imaging
MeSH Terms: conditions — CADASIL

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CADASIL cohort
- Control Cohort

SUMMARY:
The aim of this project is to establish an Australian cohort of patients diagnosed with Cerebral Autosomal Dominant Arteriopathy with Subcortical Infarcts and Leukoencephalopathy (CADASIL). This study will examine the clinical features and longitudinal course of CADASIL. Outcome measures include neuropsychological profile, neuroimaging, genetics, blood biomarkers, and retinal imaging.

DETAILED DESCRIPTION:
Using clinical examination, questionnaires, neuropsychological evaluation, brain MRI, blood sample evaluation and retinal imaging, we aim to characterise the clinical profile and progression of CADASIL in an Australian cohort.

This is multi-centre observational cohort study currently based at six sites (clinics, hospitals and universities) across three states in Australia (New South Wales, Victoria and Queensland). The multidisciplinary team aims to be the first to develop an Australian cohort of CADASIL which will contribute to global efforts and understanding of the disease.

ELIGIBILITY:
Inclusion criteria:

1. Adults ≥18 years old
2. Ability to provide written informed consent

   * A large-print version is available for individuals with visual impairment
   * An easy-to-read version is available for individuals with cognitive difficulties who may require extra support
3. Ability to attend a testing site
4. Ability to complete minimum dataset (medical examination and medical history questionnaire, blood test to determine genetic status and a short (20 minute) neuropsychology assessment).
5. CADASIL participants according to one of the following categories:

   1. confirmed diagnosis via genetic testing (NOTCH3 pathogenic variant), OR
   2. suspected diagnosis based on medical history and brain MRI, OR
   3. first degree relative of participant who is positive for NOTCH3 pathogenic variant

OR 6. Unrelated individual who is negative for the NOTCH3 pathogenic variant, and has no cognitive complaints (i.e. control participant)

Exclusion criteria:

1. Significant cognitive impairment leading to an inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with CADASIL confirmed by genetic testing, suspected due to clinical symptoms, or family history of CADASIL.
  Control cohort will be negative for the NOTCH3 pathogenic variant and have no cognitive complaints
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-11-25 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Online Medical Questionnaire | Baseline, Year 1, Year 2, Year 3, Year 4
  Includes questions on participant's medical history (CADASIL and other), family history, and medication use. Outcome will be used to inform clinical profile
Weight and height will be combined to report BMI in kg/m^2 | Baseline, Year 1, Year 2, Year 3, Year 4
  Participants will undergo structured physical examination which will provide further details on their clinical profile.
Blood Pressure | Baseline, Year 1, Year 2, Year 3, Year 4
  Participants will undergo structured physical examination which will provide further details on their clinical profile. Systolic/diastolic blood pressure will be recorded 3 times during the physical examination
Modified Rankin Scale (mRS) | Baseline, Year 1, Year 2, Year 3, Year 4
  Participants will undergo structured physical examination which will provide further details on their clinical profile. Scale from 0-5 (0 no symptoms, 5 severe disability)
National Institute of Health Stroke Scale (NIHSS) | Baseline, Year 1, Year 2, Year 3, Year 4
  Participants will undergo structured physical examination which will provide further details on their clinical profile. Individual items (11) relating to stroke symptoms and disability, for each item 0 indicates normal.
Alphabet required for Trail Making A/B | Baseline, Year 1, Year 2, Year 3, Year 4
  As part of the neuropsychological battery, participants will need to complete the alphabet to inform ability to complete Trail Making tests A and B. These indicate executive function
Montreal Cognitive Assessment (MoCA) | Baseline, Year 1, Year 2, Year 3, Year 4
  As part of the neuropsychological battery, participants will complete the MoCA to provide a measure of global cognitive function
Category Fluency (animals) | Baseline, Year 1, Year 2, Year 3, Year 4
  As part of the neuropsychological battery, participants will complete Category Fluency to provide a measure of processing speed
Digit Span Backwards (WAIS-IV) | Baseline, Year 1, Year 2, Year 3, Year 4
  As part of the neuropsychological battery, participants will complete digit span backwards to provide a measure of executive function
National Institute of Health Computerised Toolbox (NIHCTB) | Baseline, Year 1, Year 2, Year 3, Year 4
  As part of the neuropsychological battery, participants will complete the NIHCTB to provide measures of global function
Letter Fluency (FAS) | Baseline, Year 1, Year 2, Year 3, Year 4
  As part of the neuropsychological battery, participants will complete the FAS to provide measures of executive function
Rey Auditory Verbal Learning Test (RAVLT) | Baseline, Year 1, Year 2, Year 3, Year 4
  As part of the neuropsychological battery, participants will complete the RAVLT to provide measures of learning and memory
Brain MRI scan (total scan time 60 mins)- includes T1 weighted imaging | Baseline, Year 3
  To assess brain morphology
Brain MRI scan (total scan time 60 mins)- includes T2-weighted fluid attenuated inversion recovery (FLAIR) imaging | Baseline, Year 3
  Combined with T1 outcome to assess brain morphology
Brain MRI scan (total scan time 60 mins)- includes susceptibility-weighted MRI | Baseline, Year 3
  Assesses cerebral microbleeds. Signal magnitude will be processed to estimate signal decay time (i.e., T2* maps), which reflect compartmentalisation of magnetised tissue constituents (iron, calcium) [22]. Signal phase will be processed for quantitative susceptibility mapping.
Brain MRI scan (total scan time 60 mins)- includes multi-shell diffusion weighted MRI | Baseline, Year 3
  Measures of brain white matter microstructural integrity, such as fractional anisotropy and mean diffusivity, will be calculated using tensor models. Fixel-based analyses of fibre density and cross-section will also be performed. Markers of cerebrovascular diseases derived from diffusion data, such as Peak width of Skeletonised Mean Diffusivity (PSMD), will be calculated. Structural connectivity will also be examined.
Brain MRI scan (total scan time 60 mins)- includes pseudo-continuous arterial spin labelling (PCASL) perfusion imaging with multiple post-labelling delays. | Baseline, Year 3
  Used to assess quantitative cerebral blood flow and arterial transit time.
Brain MRI scan (total scan time 60 mins)- includes resting-state blood oxygenation level dependent (BOLD) imaging. | Baseline, Year 3
  Used to assess brain functional activity and amplitude of low-frequency fluctuations which embeds signal of cerebrovascular reactivity. For sites with available capnography monitors, participants' end-tidal carbon dioxide concentrations will be recorded during acquiring resting-state BOLD data for more accurate quantification of cerebrovascular reactivity

SECONDARY OUTCOMES:
Blood biochemistry | Baseline, Year 3
  Analysed by local pathology lab to indicate clinical profile. Measures will include fasting glucose, HbA1c, lipids, C-reactive protein, creatinine, vit D and liver function tests.
Ocular Questionnaire | Baseline, Year 3
  Includes questions regarding vision ability and ocular symptoms, and history
Genetic Profile | Baseline
  Genetic testing for NOTCH3 variants as well as potentially modifying genes
Instrumental Activities of Daily Living Scale (IADL) | Baseline
  Completed online, 8 items to assess daily living skills in older adults. Outcome will be used to inform clinical profile
Quality of Life Scale (EQ-5D-5L) | Baseline
  Completed online, 6 items to assess mobility, self-care, activities, pain/discomfort, anxiety/depression. Outcome will be used to inform clinical profile
STOP-BANG Sleep Questionnaire | Baseline
  Completed online, 8 items to assess Obstructive Sleep Apnoea risk. Outcome will be used to inform clinical profile
PROMIS Sleep Disturbance | Baseline
  Completed online, 8 items to assess sleep quality. Outcome will be used to inform clinical profile
Apathy Evaluation Scale (AES) | Baseline
  Completed online, 18 items to assess apathy by goal-directed behaviour, goal-related cognition, and goal-related emotional responses. Outcome will be used to inform clinical profile
Multidimensional Fatigue Inventory (MFI) | Baseline
  Completed online, 20 items to assess physical and mental fatigue and motivation. Outcome will be used to inform clinical profile
Patient Health Questionnaire-9 (PHQ-9) | Baseline
  Completed online, 9 items to assess depression symptoms and severity. Outcome will be used to inform clinical profile
Hospital Anxiety and Depression Scale (HADS) | Baseline
  Completed online, includes 14 items to assess non-physical symptoms of anxiety and depression. Outcome will be used to inform clinical profile
Study Partner Apathy Evaluation Scale (AES) | Baseline
  Completed online by nominated study partner (someone who knows the participant well e.g. spouse, carer, friend etc). Inform's participant's apathy by goal-directed behaviour, goal-related cognition, and goal-related emotional responses
Study Partner Instrumental Activities of Daily Living Scale (IADL) | Baseline
  Completed online by nominated study partner (someone who knows the participant well e.g. spouse, carer, friend etc). 8 items to assess daily living skills in older adults. Outcome will be used to inform participant's clinical profile
Neuropsychiatric Inventory (NPI-Q) | Baseline
  Completed online by nominated study partner (someone who knows the participant well e.g. spouse, carer, friend etc). 12 domains, approx. 100 questions. Used to inform psychopathology in participants
Blood Omic investigation | Baseline and year 3
  Blood tubes will be transported to the University of New South Wales for genomics, proteomics, lipidomics, and epigenomics analysis
Ocular Assessment-Visual Acuity | Baseline and year 3
  a measure of the vision function using high contrast letters will be performed with standardised vision charts at distance and at near.
Ocular Assessment- Contrast Sensitivity | Baseline and year 3
  A measure of vision function, relating to the ability to distinguish between an object and the background behind it.
Ocular Assessment- Stereopsis | Baseline and year 3
  The perception of depth will be measured using a stereo acuity instrument by viewing a series of stereograms.
Ocular Assessment- Slit-lamp examination | Baseline and year 3
  Involves viewing of the ocular structures using a slit-lamp illumination system and biomicroscope viewing system. The slit-lamp examination will be conducted by a trained observer and will allow identification of ocular media opacities, abnormalities of the eye lids, tear film and anterior structures.
Ocular Assessment- Standard automated perimetry | Baseline and year 3
  A measure of the sensitivity of the visual field.
Ocular Assessment- Intraocular pressure | Baseline and year 3
  A measure of the pressure within the eye.
Ocular Assessment- Fundus imaging (requires pupil dilation using tropicamide 0.5 or 1.0% eye drops | Baseline and year 3
  Used to visualise the back of the eye
Ocular Assessment- Optical Coherence Tomography (OCT) and OCT-Angiography | Baseline and year 3
  Used to visualise the back of the eye in retinal layers, and the retinal vessels

CONTACTS AND LOCATIONS:
Overall Officials: Perminder S Sachdev, MBBS, MD, PhD, FRANZCP, FAAHMS, Principal Investigator — University of New South Wales
Locations (5):
- Australia (5):
  - John Hunter Hospital, Newcastle, New South Wales
  - Prince of Wales Hospital, Sydney, New South Wales
  - University of New South Wales, Sydney, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Royal Melbourne Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Undecided